CLINICAL TRIAL: NCT03935087
Title: Improvement of Left Ventricular Ejection Fraction in ICD Patients Undergoing Therapy With Sacubitril/Valsartan and Potential Impact on ICD Implant Rates for Primary Prevention of Sudden Cardiac Death (SAVE-ICD)
Brief Title: Improvement of Left Ventricular Ejection Fraction in ICD Patients Undergoing Therapy With Sacubitril/Valsartan
Acronym: SAVE-ICD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Other Study IDs: SAVE-ICD
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: two-dimensional echocardiogram — two-dimensional echocardiogram with evaluation of left ventricle volumes and of left ventricular ejection fraction

SUMMARY:
The study is aimed to evaluate the improvement of the left ventricular volumes and of the left ventricular ejection fraction in a population of ICD patients with heart failure and left ventricle systolic dysfunction undergoing therapy with Sacubitril/Valsartan (according to current Guidelines), during a 6-month follow-up.

DETAILED DESCRIPTION:
Consecutive, unselected patients with heart failure and left ventricle systolic dysfunction, carrying a single-chamber or a bicameral implantable cardioverter defibrillator (ICD) for primary prevention of sudden death, undergoing therapy with Sacubitril/Valsartan (according to current Guidelines) will be enrolled in the study. A two-dimensional echocardiogram with evaluation of left ventricular end-diastolic volume, left ventricular end-systolic volume, and left ventricular ejection fraction will be performed, according to standard clinical practice, at the beginning of the observation, and at a 6-month follow-up. The improvement of the left ventricle volumes and of the left ventricular ejection fraction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* heart failure
* left ventricular systolic dysfunction
* carrying a single-chamber or a bicameral implantable cardioverter defibrillator implanted for primary prevention of sudden death
* undergoing therapy with Sacubitril/Valsartan according to current Guidelines

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure, left ventricular systolic dysfunction, carrying a single-chamber or a bicameral implantable cardioverter defibrillator implanted for primary prevention of sudden death, and undergoing therapy with Sacubitril/Valsartan according to current Guidelines
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in left ventricular ejection fraction | at enrollment and at 6 months of follow-up
  Difference between the ejection fraction observed at baseline and that observed at 6 months of follow-up

SECONDARY OUTCOMES:
Reduction in left ventricle volumes | at enrollment and at 6 months of follow-up
  Difference between the left ventricle volumes measured at baseline and those measured at 6 months of follow-up

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - "Card. G. Panico" Hospital, Tricase, Lecce
  - Federico Guerra, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna
  - AO Pugliese-Ciaccio, Catanzaro
  - Monaldi Hospital, Napoli
  - AOU "Maggiore della Carità", Novara